CLINICAL TRIAL: NCT02439749
Title: Global Clinical Study of Renal Denervation With the Symplicity Spyral™ Multi-electrode Renal Denervation System in Patients With Uncontrolled Hypertension in the Absence of Antihypertensive Medications (SPYRAL PIVOTAL - SPYRAL HTN-OFF MED)
Brief Title: SPYRAL PIVOTAL - SPYRAL HTN-OFF MED Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPYRAL HTN-OFF MED
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Results first posted 2021-05-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases
Keywords: Uncontrolled hypertension; Renal denervation
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- Renal Denervation (Experimental): Renal angiography and Renal Denervation (Symplicity Spyral™ multi-electrode renal denervation system)
  Interventions: Device: Symplicity Spyral™ multi-electrode renal denervation system
- Sham Procedure (Sham Comparator): Renal angiography
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Device: Symplicity Spyral™ multi-electrode renal denervation system — After a renal angiography according to standard procedures, subjects remain blinded and are immediately treated with the renal denervation procedure after randomization.
  Other Names: Renal angiography; Renal Denervation
  Arms: Renal Denervation
Procedure: Sham Procedure — After a renal angiography according to standard procedures, subjects remain blinded and remain on the catheterization lab table for at least 20 minutes prior to introducer sheath removal.
  Other Names: Renal angiography
  Arms: Sham Procedure

SUMMARY:
The purpose of this study is to test the hypothesis that renal denervation decreases blood pressure and is safe when studied in the absence of antihypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

* Individual has office systolic blood pressure (SBP) ≥ 150 mmHg and <180 mmHg and a diastolic blood pressure (DBP) ≥ 90 mmHg after being off medications.
* Individual has 24-hour Ambulatory Blood Pressure Monitoring (ABPM) average SBP ≥ 140 mmHg and < 170 mmHg.
* Individual is willing to discontinue current antihypertensive medications.

Exclusion Criteria:

* Individual lacks appropriate renal artery anatomy.
* Individual has estimated glomerular filtration rate (eGFR) of <45.
* Individual has type 1 diabetes mellitus or poorly-controlled type 2 diabetes mellitus.
* Individual has one or more episodes of orthostatic hypotension.
* Individual requires chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea.
* Individual has primary pulmonary hypertension.
* Individual is pregnant, nursing or planning to become pregnant.
* Individual has frequent intermittent or chronic pain that results in treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) for two or more days per week over the month prior to enrollment.
* Individual has stable or unstable angina within 3 months of enrollment, myocardial infarction within 3 months of enrollment; heart failure, cerebrovascular accident or transient ischemic attack, or atrial fibrillation at any time.
* Individual works night shifts.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Townsend, MD, Principal Investigator — University of Pennsylvania; David Kandzari, MD, Principal Investigator — Piedmont Hospital; Michael Böhm, MD, Principal Investigator — Universitätskliniken des Saarlandes; Kazuomi Kario, MD, Principal Investigator — Jichi Medical University
Locations (47):
- United States (30):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Honor Health Research Institute, Scottsdale, Arizona
  - Kaiser Permanente LA Medical Center, Los Angeles, California
  - Stanford Hospital and Clinics, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Kentucky, Lexington, Kentucky
  - St Joseph Mercy Oakland, Pontiac, Michigan
  - Providence Hospital, Southfield, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Cardiology Associates Research LLC, Tupelo, Mississippi
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - PinnacleHealth Cardiovascular Institute, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - Charleston Area Medical Center, Charleston, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Alfred Hospital, Melbourne, Victoria, Australia
- Klinikum Wels-Grieskirchen, Wels, Austria
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Institut de cardiologie de Montréal / Montreal Heart Institute, Montreal, Quebec
- Germany (5):
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen GmbH, Bad Krozingen
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum des Saarlandes, Homburg
  - Herzzentrum Leipzig, Universitätsklinik, Leipzig
  - Sana Kliniken Lübeck, Lübeck
- Greece (2):
  - Hippokration General Hospital of Athens, Athens
  - University General Hospital of Thessaloniki (AHEPA), Thessaloniki
- Galway University Hospital, Galway, Ireland
- Japan (2):
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Mitsui Memorial Hospital, Chiyoda City, Tokyo
- United Kingdom (3):
  - Cardiff and Vale University Health Board - University Hospital of Wales, Cardiff
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Derived] Weber MA, Schmieder RE, Kandzari DE, Townsend RR, Mahfoud F, Tsioufis K, Kario K, Pocock S, Tatakis F, Ewen S, Choi JW, East C, Lee DP, Ma A, Cohen DL, Wilensky R, Devireddy CM, Lea JP, Schmid A, Fahy M, Bohm M. Hypertension urgencies in the SPYRAL HTN-OFF MED Pivotal trial. Clin Res Cardiol. 2022 Nov;111(11):1269-1275. doi: 10.1007/s00392-022-02064-5. Epub 2022 Jul 19. PMID 35852582
- [Derived] Bohm M, Tsioufis K, Kandzari DE, Kario K, Weber MA, Schmieder RE, Townsend RR, Kulenthiran S, Ukena C, Pocock S, Ewen S, Weil J, Fahy M, Mahfoud F. Effect of Heart Rate on the Outcome of Renal Denervation in Patients With Uncontrolled Hypertension. J Am Coll Cardiol. 2021 Sep 7;78(10):1028-1038. doi: 10.1016/j.jacc.2021.06.044. PMID 34474735
- [Derived] Mahfoud F, Townsend RR, Kandzari DE, Kario K, Schmieder RE, Tsioufis K, Pocock S, David S, Patel K, Rao A, Walton A, Bloom JE, Weber T, Suppan M, Lauder L, Cohen SA, McKenna P, Fahy M, Bohm M, Weber MA. Changes in Plasma Renin Activity After Renal Artery Sympathetic Denervation. J Am Coll Cardiol. 2021 Jun 15;77(23):2909-2919. doi: 10.1016/j.jacc.2021.04.044. Epub 2021 May 3. PMID 33957242
- [Derived] Bohm M, Kario K, Kandzari DE, Mahfoud F, Weber MA, Schmieder RE, Tsioufis K, Pocock S, Konstantinidis D, Choi JW, East C, Lee DP, Ma A, Ewen S, Cohen DL, Wilensky R, Devireddy CM, Lea J, Schmid A, Weil J, Agdirlioglu T, Reedus D, Jefferson BK, Reyes D, D'Souza R, Sharp ASP, Sharif F, Fahy M, DeBruin V, Cohen SA, Brar S, Townsend RR; SPYRAL HTN-OFF MED Pivotal Investigators. Efficacy of catheter-based renal denervation in the absence of antihypertensive medications (SPYRAL HTN-OFF MED Pivotal): a multicentre, randomised, sham-controlled trial. Lancet. 2020 May 2;395(10234):1444-1451. doi: 10.1016/S0140-6736(20)30554-7. Epub 2020 Mar 29. PMID 32234534
- [Derived] Bohm M, Townsend RR, Kario K, Kandzari D, Mahfoud F, Weber MA, Schmieder RE, Tsioufis K, Hickey GL, Fahy M, DeBruin V, Brar S, Pocock S. Rationale and design of two randomized sham-controlled trials of catheter-based renal denervation in subjects with uncontrolled hypertension in the absence (SPYRAL HTN-OFF MED Pivotal) and presence (SPYRAL HTN-ON MED Expansion) of antihypertensive medications: a novel approach using Bayesian design. Clin Res Cardiol. 2020 Mar;109(3):289-302. doi: 10.1007/s00392-020-01595-z. Epub 2020 Feb 7. PMID 32034481
- [Derived] Townsend RR, Mahfoud F, Kandzari DE, Kario K, Pocock S, Weber MA, Ewen S, Tsioufis K, Tousoulis D, Sharp ASP, Watkinson AF, Schmieder RE, Schmid A, Choi JW, East C, Walton A, Hopper I, Cohen DL, Wilensky R, Lee DP, Ma A, Devireddy CM, Lea JP, Lurz PC, Fengler K, Davies J, Chapman N, Cohen SA, DeBruin V, Fahy M, Jones DE, Rothman M, Bohm M; SPYRAL HTN-OFF MED trial investigators*. Catheter-based renal denervation in patients with uncontrolled hypertension in the absence of antihypertensive medications (SPYRAL HTN-OFF MED): a randomised, sham-controlled, proof-of-concept trial. Lancet. 2017 Nov 11;390(10108):2160-2170. doi: 10.1016/S0140-6736(17)32281-X. Epub 2017 Aug 28. PMID 28859944
- [Derived] Kandzari DE, Kario K, Mahfoud F, Cohen SA, Pilcher G, Pocock S, Townsend R, Weber MA, Bohm M. The SPYRAL HTN Global Clinical Trial Program: Rationale and design for studies of renal denervation in the absence (SPYRAL HTN OFF-MED) and presence (SPYRAL HTN ON-MED) of antihypertensive medications. Am Heart J. 2016 Jan;171(1):82-91. doi: 10.1016/j.ahj.2015.08.021. Epub 2015 Sep 11. PMID 26699604

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Renal Denervation | Sham Procedure
Started | 182 | 184
Completed | 153 | 147
Not Completed | 29 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Renal Denervation | Sham Procedure | Total
Number analyzed (Participants) | 182 | 184 | 366
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 158 | 167 | 325
  >=65 years | 24 | 17 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10.8) | 52.7 (10.1) | 52.6 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 56 | 121
  Male | 117 | 128 | 245
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 32 | 69
  White | 56 | 60 | 116
  Japanese from Japan | 3 | 2 | 5
  Other | 1 | 1 | 2
  Unknown or Not Reported | 78 | 87 | 165
Region of Enrollment [Number; unit: participants]
  Greece | 28 | 30 | 58
  Canada | 3 | 2 | 5
  Austria | 3 | 4 | 7
  United States | 91 | 85 | 176
  Japan | 3 | 2 | 5
  Ireland | 7 | 7 | 14
  United Kingdom | 6 | 10 | 16
  Australia | 7 | 6 | 13
  Germany | 34 | 38 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Events (MAE) Defined as a Composite of Events.
Description: All-cause mortality End-stage Renal Disease (ESRD) Significant embolic event resulting in end-organ damage Renal artery perforation requiring intervention Renal artery dissection requiring intervention Vascular complications Hospitalization for hypertensive crisis not related to confirmed non-adherence with medications or the protocol New renal artery stenosis >70% (6 months for new renal artery stenosis)
Time Frame: From baseline to 1 month post-procedure (6 months for new renal artery stenosis)
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 0

2. Primary Outcome: Baseline Adjusted Change (Using Analysis of Covariance) in Systolic Blood Pressure as Measured by 24-hour Ambulatory Blood Pressure Monitoring
Description: The outcome measure is the change in ambulatory systolic blood pressure from baseline to 3-month. The unadjusted treatment difference between renal denervation and sham control groups is -3.9 mmHg. The baseline adjusted treatment difference is -3.9 mmHg.
Time Frame: From baseline to 3 months post-procedure
Population: The number of participants analyzed reflects the number of subjects within each treatment arm who have data available for outcome measure analysis. This number can be variable from the number of subjects in each treatment arm at study start.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 153 | 147
mmHg | -4.5 (10.8) | -0.6 (8.7)

3. Secondary Outcome: Number of Participants With Significant Embolic Event Resulting in End-organ Damage
Description: Significant embolic event resulting in end-organ damage (e.g. kidney/bowel infarct, lower extremity ulceration or gangrene, or doubling of serum creatinine documented by at least two measurements at least 21 days apart)
Time Frame: From baseline to 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Renal Artery Perforation Requiring Intervention
Description: Renal artery perforation requiring intervention
Time Frame: From baseline to 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 0

5. Secondary Outcome: Renal Artery Dissection
Description: Number of Participants with Renal artery dissection requiring intervention
Time Frame: From baseline to 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Vascular Complications
Description: Vascular complications (e.g., clinically significant groin hematoma, arteriovenous fistula, pseudoaneurysm, excessive bleeding) requiring surgical repair, interventional procedure, thrombin injection, or blood transfusion (requiring more than 2 units of packed red blood cells within any 24 hour period during the first 7 days post renal denervation procedure).
Time Frame: From baseline to 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 1

7. Secondary Outcome: Number of Participants With End-stage Renal Disease
Description: defined as two or more eGFR measurements < 15 mL/min/1.73m2 at least 21 days apart and requiring dialysis for one of more of the following:
  * Volume management refractory to diuretics
  * Hyperkalemia unmanageable by diet and diuretics
  * Acidosis bicarbonate <18 unmanageable with HCO3 supplements
  * Symptoms of uremia, nausea, vomiting
Time Frame: From baseline to 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Decline in eGFR
Description: ≥40% decline in eGFR
Time Frame: From baseline to 1 month post-procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 171 | 170
Participants | 0 | 0

9. Secondary Outcome: Myocardial Infarction
Description: Number of Participants with New myocardial infarction
Time Frame: From baseline to 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 0

10. Secondary Outcome: New Stroke
Description: Number of Participants with New stroke
Time Frame: From baseline to 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Renal Artery Re-intervention
Description: Renal artery re-intervention
Time Frame: From baseline to 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Major Bleeding According to TIMI Definition
Description: Major bleeding according to TIMI definition (i.e. intracranial hemorrhage, ≥5g/dl decrease in hemoglobin concentration, a ≥15% absolute decrease in hematocrit, or death due to bleeding within 7 days of the procedure).
Time Frame: From baseline to 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Increase in Serum Creatinine
Description: Increase in serum creatinine > 50% from screening visit 2.
Time Frame: From baseline to 1 month post-procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 171 | 170
Participants | 1 | 0

14. Secondary Outcome: Number of Participants With Hospitalization for Hypertensive Crisis With Medications or the Protocol
Description: Hospitalization for hypertensive crisis not related to confirmed non-adherence with medications or the protocol.
Time Frame: From baseline to 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 182 | 184
Participants | 0 | 0

15. Secondary Outcome: Change in Office Systolic Blood Pressure
Description: Change in office systolic blood pressure from baseline (Screening Visit 2) to 1-month
Time Frame: From baseline to 1 month post procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 170 | 169
mmHg | -10.2 (14.0) | -5.7 (11.8)

16. Secondary Outcome: Change in Office Diastolic Blood Pressure
Description: Change in office diastolic blood pressure from baseline (Screening Visit 2)
Time Frame: From baseline to 1 month post procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 170 | 169
mmHg | -5.3 (8.3) | -2.9 (7.6)

17. Secondary Outcome: Number of Participants Achieving Target Office Systolic Blood Pressure
Description: Incidence of achieving target office systolic blood pressure (SBP <140 mmHg)
Time Frame: From baseline to 1 month post procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 170 | 169
Participants | 32 | 11

18. Secondary Outcome: Baseline Adjusted Change (Using Analysis of Covariance) in Office Systolic Blood Pressure
Description: The outcome measure is the change in office systolic blood pressure from baseline to 3-month. The unadjusted treatment difference between renal denervation and sham control groups is -7.0 mmHg. The baseline adjusted treatment difference is -6.9 mmHg.
Time Frame: From baseline to 3 months post-procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 170 | 164
mmHg | -9.4 (14.8) | -2.3 (12.7)

19. Secondary Outcome: Number of Participants With All-cause Mortality
Description: All-cause mortality
Time Frame: From baseline to 3 months post-procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 181 | 184
Participants | 0 | 0

20. Secondary Outcome: Number of Participants With ≥40% Decline in eGFR
Description: ≥40% Decline in eGFR
Time Frame: From baseline to 3 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 165 | 149
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With End-Stage Renal Disease (ESRD)
Description: as for outcome 7
Time Frame: From baseline to 3 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 181 | 184
Participants | 0 | 0

22. Secondary Outcome: Number of Participants With New Myocardial Infarction
Description: New Myocardial Infarction
Time Frame: From baseline to 3 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 181 | 184
Participants | 0 | 0

23. Secondary Outcome: New Stroke
Description: Number of Participants with New Stroke
Time Frame: From baseline to 3 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 181 | 184
Participants | 0 | 1

24. Secondary Outcome: Number of Participants With Renal Artery Re-intervention
Description: Renal Artery Re-intervention
Time Frame: From baseline to 3 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 181 | 184
Participants | 0 | 0

25. Secondary Outcome: Number of Participants With Major Bleeding According to TIMI Definition
Description: as for outcome 12
Time Frame: From baseline to 3 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 181 | 184
Participants | 0 | 0

26. Secondary Outcome: Increase in Serum Creatinine
Description: Number of Participants with Increase in Serum Creatinine > 50% from screening visit 2.
Time Frame: From baseline to 3 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 165 | 149
Participants | 0 | 0

27. Secondary Outcome: Number of Participants With Hospitalization for Hypertensive Crisis
Description: Hospitalization for Hypertensive Crisis Not Related to Confirmed Nonadherence With Medications or the Protocol
Time Frame: From baseline to 3 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 181 | 184
Participants | 1 | 0

28. Secondary Outcome: Change in Diastolic Blood Pressure as Measured by 24-hour ABPM
Description: Change in diastolic blood pressure from baseline (screening visit 2) to 3-month as measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM).
Time Frame: From baseline to 3 months post procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 153 | 147
mmHg | -3.5 (6.7) | -0.8 (5.7)
Statistical Analysis 1: Comparison: Renal Denervation vs Sham Procedure; Test type: Superiority; p < 0.001, ANCOVA — p<0.05 required for significance

29. Secondary Outcome: Change in Office Diastolic Blood Pressure
Description: Change in Office Diastolic Blood Pressure From Baseline (Screening Visit 2) to 3-months
Time Frame: From baseline to 3 months post procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 170 | 164
mmHg | -5.0 (8.3) | -1.0 (8.0)

30. Secondary Outcome: Number of Participants Achieving Target Office Systolic Blood Pressure
Description: Incidence of Achieving Target Office Systolic Blood Pressure (SBP <140 mmHg)
Time Frame: From baseline to 3 months post procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 170 | 164
Participants | 27 | 12

31. Secondary Outcome: Number of Participants With New Renal Artery Stenosis > 70%
Description: Confirmed by angiography and as determined by the angiographic core laboratory.
Time Frame: From baseline to 6 month post-procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 163 | 125
Participants | 0 | 0

32. Secondary Outcome: Change in Systolic Blood Pressure as Measured by 24-hour ABPM
Time Frame: From baseline to 36 month post-procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 127 | 39
mmHg | -16.2 (14.6) | -22.0 (13.3)
Statistical Analysis 1: Comparison: Renal Denervation vs Sham Procedure; Test type: Superiority; p = 0.026, ANCOVA — p<0.05 required for significance

33. Secondary Outcome: Change in Diastolic Blood Pressure as Measured by 24-hour ABPM
Description: Change in diastolic blood pressure as measured by 24-hour ABPM
Time Frame: From baseline to 36 months post-procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 127 | 39
mmHg | -11.7 (9.6) | -15.0 (8.0)
Statistical Analysis 1: Comparison: Renal Denervation vs Sham Procedure; Test type: Superiority; p = 0.052, ANCOVA — p<0.05 required for significance

34. Secondary Outcome: Change in Office Systolic Blood Pressure
Description: Change in Office Systiloc Blood Pressure From Baseline (Screening Visit 2) to 36 months.
Time Frame: From baseline to 36 months post procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 154 | 47
mmHg | -21.9 (15.5) | -26.4 (12.8)
Statistical Analysis 1: Comparison: Renal Denervation vs Sham Procedure; Test type: Superiority; p = 0.070, ANCOVA — p<0.05 required for significance

35. Secondary Outcome: Change in Office Diastolic Blood Pressure
Description: Change in office diastolic blood pressure
Time Frame: From baseline to 36 months post-procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 154 | 47
mmHg | -10.8 (10.4) | -15.4 (10.8)
Statistical Analysis 1: Comparison: Renal Denervation vs Sham Procedure; Test type: Superiority; p = 0.009, ANCOVA — p=<0.05 required for significance

36. Secondary Outcome: Number of Participants With Incidence of Achieving Target Office Systolic Blood Pressure (SBP <140) mmHg)
Time Frame: From baseline to 36 months post-procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 154 | 47
Participants | 70 | 33

37. Secondary Outcome: Number of Participants With All-cause Mortality
Time Frame: From baseline to 36 months post-randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 166 | 104
Participants | 0 | 1

38. Secondary Outcome: Number of Participants With End-Stage Renal Disease (ESRD)
Description: as for outcome 7
Time Frame: From baseline to 36 months post randomization
Population: The number of participants analyzed reflects the number of subjects within each treatment arm who have data available for outcome measure analysis. This number can be variable from the number of subjects in each treatment are at study start.
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 166 | 104
Participants | 0 | 0

39. Secondary Outcome: Number of Participants With ≥40% Decline in eGFR
Description: ≥40% Decline in eGFR
Time Frame: From baseline to 36 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 144 | 40
Participants | 1 | 0

40. Secondary Outcome: Number of Participants With New Myocardial Infarction
Description: New Myocardial Infarction
Time Frame: From baseline to 36 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 166 | 104
Participants | 0 | 0

41. Secondary Outcome: Number of Participants With New Stroke
Description: New Stroke
Time Frame: From baseline to 36 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 166 | 104
Participants | 0 | 3

42. Secondary Outcome: Number of Participants With Renal Artery Re-intervention
Description: Renal Artery Re-intervention
Time Frame: From baseline to 36 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 166 | 104
Participants | 0 | 0

43. Secondary Outcome: Number of Participants With Major Bleeding According to TIMI Definition
Description: as for outcome 12
Time Frame: From baseline to 36 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 166 | 104
Participants | 0 | 2

44. Secondary Outcome: Number of Participants With an Increase in Serum Creatinine
Description: Number of Participants with Increase in Serum Creatinine > 50% from screening visit 2.
Time Frame: From baseline to 36 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 144 | 40
Participants | 1 | 0

45. Secondary Outcome: Number of Participants With New Renal Artery Stenosis > 70%
Description: Confirmed by angiography and as determined by the angiographic core laboratory.
Time Frame: From baseline to 36 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 166 | 104
Participants | 0 | 0

46. Secondary Outcome: Number of Participants With Hospitalization for Hypertensive Crisis
Description: Hospitalization for hypertensive crisis not related to confirmed non-adherence with medications orthe protocol
Time Frame: From baseline to 36 months post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 166 | 104
Participants | 1 | 2

47. Other Pre Specified Outcome: Antihypertensive Medication Burden to 36-months
Description: Based on the prescribed medications reported, medication burden was calculated using Medication Index 2 score which is a composite index based on the doses of antihypertensive medications multiplied by the number of medications prescribed; all classes (ACE/ARB, calcium channel blockers, etc.) were considered equivalent in potency. Higher score indicates higher dosages being prescribed over the standard dose.
  There are no clinically established thresholds.
Time Frame: From baseline to 36 months post-procedure
Population: The number of participants analyzed reflects the number of subjects with prescribed medications reported.
Measure: Mean (Standard Deviation); unit: Medication Index 2 Score
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 165 | 54
Medication Index 2 Score | 2.09 (2.40) | 3.20 (3.60)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Serious Adverse Events were monitored/assessed from subject enrollment (consent) through study exit (up to 36 Months Post Procedure) while Other Adverse Events were monitored/assessed from subject enrollment (consent) through 12-month visits.
Description: The number of participants analyzed reflects the number of subjects within each treatment arm who have data available for outcome measure analysis. This number can be variable from the number of subjects in each treatment arm at study start.
Arm/Group | Renal Denervation | Sham Procedure
All-Cause Mortality (participants affected / at risk) | 1/182 | 2/184
Serious Adverse Events (participants affected / at risk) | 38/182 | 36/184
Other Adverse Events (participants affected / at risk) | 149/182 | 155/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Denervation (N=182) | Sham Procedure (N=184)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Basal Ganglia Hemorrage (Nervous system disorders) | 0 (0) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal Uterine Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0)
Mast Cell Activation Syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Superventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Mucosal Lesion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic Shock (Immune system disorders) | 1 (1) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Localized Infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis Externa (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) — General Disorders And Administration Site Conditions
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) — General Disorders And Administration Site Conditions
Pyrexia (General disorders) | 1 (1) | 0 (0) — General Disorders And Administration Site Conditions
Subcutaneous Abscess (Infections and infestations) | 1 (1) | 0 (0)
Systemic Candida (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shoulder Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Arthrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Access Site Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiac Stress Test Abnormal (Investigations) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Melanoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Focal Dyscognitive Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhagic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial Pressure Increased (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Primary Headache Associated With Sexual Activity (Nervous system disorders) | 0 (0) | 1 (1)
Thalamic Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 1 (1)
Ruptured Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic Organ Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Obstructive Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Cataract Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Percutaneous Coronary Intervention (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Emergency (Vascular disorders) | 0 (0) | 0 (0)
Varicose Vein (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Denervation (N=182) | Sham Procedure (N=184)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mast Cell Activation Syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Aortic Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bundle Branch Block Left (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Left Ventricular Hypertrophy (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 2 (2)
Sinus Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular Tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goiter (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0)
Conjunctival Hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Floppy Eyelid Syndrome (Eye disorders) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Ocular Hyperemia (Eye disorders) | 0 (0) | 1 (1)
Optic Nerve Disorder (Eye disorders) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 2 (2) | 2 (2)
Visual Impairment (Eye disorders) | 2 (2) | 4 (4)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal Mass (Gastrointestinal disorders) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Angular Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Adverse Drug Reaction (General disorders) | 2 (2) | 0 (0) — General Disorders and Administration Site Conditions
Asthenia (General disorders) | 1 (1) | 1 (1) — General Disorders and Administration Site Conditions
Axillary Pain (General disorders) | 0 (0) | 1 (1) — General Disorders and Administration Site Conditions
Chest Discomfort (General disorders) | 3 (3) | 2 (2) — General Disorders and Administration Site Conditions
Chest Pain (General disorders) | 4 (4) | 5 (5) — General Disorders and Administration Site Conditions
Drug Intolerance (General disorders) | 1 (1) | 1 (1) — General Disorders and Administration Site Conditions
Fatigue (General disorders) | 6 (6) | 9 (9) — General Disorders and Administration Site Conditions
Feeling Hot (General disorders) | 0 (0) | 1 (1) — General Disorders and Administration Site Conditions
Gait Disturbance (General disorders) | 0 (0) | 1 (1) — General Disorders and Administration Site Conditions
Impaired Healing (General disorders) | 0 (0) | 1 (1) — General Disorders and Administration Site Conditions
Influenza Like Illness (General disorders) | 1 (1) | 3 (3) — General Disorders and Administration Site Conditions
Malaise (General disorders) | 0 (0) | 1 (1) — General Disorders and Administration Site Conditions
Medical Device Site Irritation (General disorders) | 0 (0) | 1 (1) — General Disorders and Administration Site Conditions
Medical Device Site Pain (General disorders) | 0 (0) | 1 (1) — General Disorders and Administration Site Conditions
Medical Device Site Pruritus (General disorders) | 0 (0) | 1 (1) — General Disorders and Administration Site Conditions
Medical Device Site Reaction (General disorders) | 0 (0) | 0 (0) — General Disorders and Administration Site Conditions
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 6 (6) — General Disorders and Administration Site Conditions
Oedema (General disorders) | 0 (0) | 0 (0) — General Disorders and Administration Site Conditions
Oedema Peripheral (General disorders) | 12 (12) | 15 (15) — General Disorders and Administration Site Conditions
Pain (General disorders) | 1 (1) | 2 (2) — General Disorders and Administration Site Conditions
Peripheral Swelling (General disorders) | 2 (2) | 5 (5) — General Disorders and Administration Site Conditions
Puncture Site Reaction (General disorders) | 1 (1) | 0 (0) — General Disorders and Administration Site Conditions
Pyrexia (General disorders) | 1 (1) | 3 (3) — General Disorders and Administration Site Conditions
Swelling (General disorders) | 0 (0) | 1 (1) — General Disorders and Administration Site Conditions
Swelling Face (General disorders) | 1 (1) | 0 (0) — General Disorders and Administration Site Conditions
Vessel Puncture Site Pain (General disorders) | 0 (0) | 1 (1) — General Disorders and Administration Site Conditions
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Contrast Media Reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 3 (3) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0)
Borrelia Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Diarrhea Infectious (Infections and infestations) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal Foot Infection (Infections and infestations) | 0 (0) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (3)
Gastrointestinal Viral Infection (Infections and infestations) | 0 (0) | 2 (2)
H1n1 Influenza (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter Gastritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes Simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 8 (8) | 6 (6)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Localized Infection (Infections and infestations) | 1 (1) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Lyme Disease (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (11) | 14 (14)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis Externa (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3) | 4 (4)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 7 (7) | 6 (6)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 5 (5)
Vaginal Infection (Infections and infestations) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Vestibular Neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns Second Degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Chemical Burn Of Skin (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Corneal Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dislocation Of Vertebra (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision Site Complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision Site Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incision Site Pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament Rupture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Muscle Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Post Procedural Hematoma (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Post Procedural Hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Site Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal Column Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic Arthrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Access Site Bruising (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 16 (16) | 22 (22)
Vascular Access Site Hemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Vascular Access Site Pain (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular Pseudoaneurysm Thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood Cholesterol Increased (Investigations) | 2 (2) | 2 (2)
Blood Creatinine Increased (Investigations) | 4 (4) | 3 (3)
Blood Glucose Increased (Investigations) | 2 (2) | 1 (1)
Blood Magnesium Decreased (Investigations) | 0 (0) | 1 (1)
Blood Potassium Decreased (Investigations) | 0 (0) | 1 (1)
Blood Pressure Abnormal (Investigations) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 5 (5) | 4 (4)
Blood Pressure Orthostatic Decreased (Investigations) | 1 (1) | 0 (0)
Blood Pressure Systolic Increased (Investigations) | 0 (0) | 4 (4)
Blood Uric Acid Increased (Investigations) | 0 (0) | 4 (4)
C-Reactive Protein Increased (Investigations) | 1 (1) | 0 (0)
Cardiac Murmur (Investigations) | 0 (0) | 1 (1)
Cardiac Stress Test Abnormal (Investigations) | 0 (0) | 1 (1)
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 2 (2)
Hemoglobin Abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0)
Lipids Increased (Investigations) | 0 (0) | 0 (0)
Occult Blood (Investigations) | 0 (0) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 1 (1) | 0 (0)
Renin Decreased (Investigations) | 1 (1) | 0 (0)
Respiratory Rate Decreased (Investigations) | 1 (1) | 0 (0)
Troponin Increased (Investigations) | 0 (0) | 1 (1)
Urine Analysis Abnormal (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypercholesterolemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insulin Resistance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 13 (13)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 8 (8)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Knee Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Tendon Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypergammaglobulinemia Benign Monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Melanoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Paraganglion Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid Tumor Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Renal Hamartoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cranial Nerve Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 15 (15) | 12 (12)
Dizziness Postural (Nervous system disorders) | 1 (1) | 4 (4)
Drug Withdrawal Headache (Nervous system disorders) | 0 (0) | 0 (0)
Electric Shock Sensation (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Essential Tremor (Nervous system disorders) | 0 (0) | 0 (0)
Focal Dyscognitive Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 32 (32) | 31 (31)
Hemorrhagic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hypoesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 3 (3)
Loss Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 8 (8)
Nerve Compression (Nervous system disorders) | 0 (0) | 1 (1)
Orthostatic Intolerance (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 2 (2)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1)
Primary Headache Associated With Sexual Activity (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 3 (3)
Tension Headache (Nervous system disorders) | 0 (0) | 1 (1)
Thalamic Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 1 (1)
Trigeminal Nerve Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Device Physical Property Issue (Product Issues) | 1 (1) | 0 (0)
Alcohol Use Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Depressed Mood (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Intrusive Thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Vomiting Psychogenic (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Renal Artery Occlusion (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Mass (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Breast Inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic Organ Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Dyspnea At Rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Dyspnea Paroxysmal Nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Obstructive Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin Discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Stress At Work (Social circumstances) | 1 (1) | 0 (0)
Facet Joint Block (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Wisdom Teeth Removal (Surgical and medical procedures) | 0 (0) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Arterial Spasm (Vascular disorders) | 1 (1) | 0 (0)
Circulatory Collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 0 (0)
Giant Cell Arteritis (Vascular disorders) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 10 (10) | 11 (11)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 3 (3)
Hypertensive Emergency (Vascular disorders) | 0 (0) | 0 (0)
Hypertensive Urgency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 6 (6) | 4 (4)
Jugular Vein Distension (Vascular disorders) | 2 (2) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Peripheral Coldness (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Venous Disease (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Systolic Hypertension (Vascular disorders) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT02439749/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT02439749/SAP_001.pdf